CLINICAL TRIAL: NCT06956924
Title: CT-Based Abdominal Aortic Calcium Score and CAD-RADS 2.0 in Elderly Chest Pain: A Cohort Study
Brief Title: Abdominal Aortic Calcium and CAD-RADS 2.0
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: liao1009_01; CMRPG8L0731 (Other Grant/Funding Number: Kaohsiung Chang-Gung Memorial Hospital)
Record Dates: First submitted 2025-04-16; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease (CAD)
Keywords: Coronary Artery Disease (CAD); Abdominal Aortic Calcium (AAC); Coronary Artery Calcium (CAC); CAD-RADS 2.0 Classification; Coronary Plaque Burden
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CCTA and Non-Enhanced Abdominal CT Scan Protocol (Experimental): CCTA was performed using a 640-slice multislice CT scanner (Canon Aquilion One Genesis, Canon Medical Systems, Japan). All participants received sublingual nitroglycerin (0.3 mg) to promote coronary vasodilation prior to imaging. The first phase involved an unenhanced, prospective electrocardiogram (ECG)-gated volume scan for CAC assessment, configured to 120 kVp and 50 mAs with a field of view (FOV) of 16 cm to ensure comprehensive cardiac coverage. Imaging was performed with a rotation time of 0.275 seconds and a slice thickness of 2 mm. Following this, an abdominal aorta scan was performed using a non-ECG-gated sequential scan mode, maintaining identical settings of 120 kVp and 2 mm slice thickness. The inferior aspect of the L5 vertebral body endplate was used as the caudal extent of the abdominal volume to be imaged, covering the iliac bifurcation of the infrarenal abdominal aorta while minimizing radiation exposure to the pelvic genital organs.
  Interventions: Diagnostic Test: CCTA

INTERVENTIONS:
Diagnostic Test: CCTA — The data acquisition protocol was tailored to each patient's heart rate and rhythm. Specifically, a prospectively ECG-triggered volume scan was used to account for heart rates and rhythms, capturing predefined scanning areas during R-R intervals, especially in instances of frequent ectopic beats or irregular heart rates noted during pre-scan ECG monitoring. Imaging system parameters included a gantry rotation time of 0.275 seconds, collimation of 0.5 mm, tube voltage settings ranging from 100 kV to 120 kV, and a tube current-time product between 200 mAs and 450 mAs, with adjustments based on the patient's BMI.

SUMMARY:
Background: Abdominal aortic calcium (AAC) is a marker of systemic atherosclerosis and may predict cardiovascular outcomes similarly to coronary artery calcium (CAC). This study evaluates the predictive efficacy of CT-based AAC scores for coronary plaque burden and stenosis using the CAD-RADS 2.0 classification system.

Methods: A prospective cohort of 68 patients (mean age 67.5 years) with chest pain underwent cardiac CT for CAC, AAC scoring, and coronary computed tomography angiography (CCTA) at Kaohsiung Chang Gung Memorial Hospital (June 2021-May 2023). AAC scores were quantified using the Agatston method across 8 cm and 5 cm aortic segments, and outcomes were analyzed based on CAD-RADS 2.0 and plaque burden classifications.

DETAILED DESCRIPTION:
Introduction Coronary artery calcium (CAC) scoring, developed and validated using computed tomography (CT), is a well-established technique for quantifying coronary atherosclerosis and assessing cardiovascular risk, thereby guiding preventive therapeutic strategies. Similarly, abdominal aortic calcium (AAC) is a biomarker indicating the degree of calcification within the abdominal aorta, reflecting systemic atherosclerosis. AAC has been shown to predict cardiovascular morbidity and mortality.

AAC can be assessed using two common methods: Kidney, Ureter, and Bladder (KUB) plain film radiography and CT. Studies have demonstrated a correlation between AAC and CAC scores, with AAC suggesting the presence of asymptomatic coronary artery disease (CAD). This highlights the potential importance of quantifying AAC in predicting CAD.

Coronary Computed Tomography Angiography (CCTA) enables direct visualization of coronary artery lumen stenosis, atherosclerotic plaque composition, and high-risk plaque features, such as low attenuation, spot calcification, positive remodeling, and the napkin ring sign. CCTA is particularly valuable in patients with stable chest pain, given its high sensitivity and specificity in detecting CAD. Furthermore, it plays a critical role in guiding decisions regarding coronary revascularization procedures. Beyond assessing coronary artery stenosis and atherosclerotic plaque characteristics, analyzing plaque volume and burden provides prognostic value in stratifying the risk of acute coronary syndrome (ACS) in patients with stable chest pain undergoing CCTA.

The Coronary Artery Disease Reporting and Data System (CAD-RADS) is a comprehensive framework designed to standardize the assessment of disease severity and guide treatment decisions in patients with CAD. Initially published in 2016, CAD-RADS employs a categorical system based on coronary artery stenosis and high-risk plaque characteristics as modifiers. The 2022 update, CAD-RADS 2.0, incorporates plaque burden as a new subclassification and assesses lesion-specific ischemia using CT fractional flow reserve (CT-FFR) or myocardial CT perfusion (CTP). CAD-RADS aims to standardize CCTA reporting and improve communication with referring physicians, including recommendations.

Previous studies have indicated a correlation between AAC and CAC, with AAC quantification linked to traditional cardiovascular risk factors and cardiovascular events. Additionally, CT-based AAC quantification can predict future cardiovascular events in asymptomatic adults. However, few studies have explored whether AAC correlates with non-calcified coronary artery plaques or the degree of coronary artery stenosis. This study aims to investigate the correlation between CT-based AAC scores and coronary plaque burden and stenosis, using the CAD-RADS 2.0 classification system.

Materials and Methods Study Population This prospective cohort study enrolled patients aged 60 years and older who presented to the cardiovascular department at Kaohsiung Chang Gung Memorial Hospital between June 2021 and May 2023. Inclusion criteria were patients with chest pain or discomfort who were scheduled to undergo cardiac CT for CAC and CCTA, as determined by the treating physician for the evaluation of CAD. Exclusion criteria included: (1) severe allergies to contrast agents, (2) metallic implants in the lumbar spine, (3) renal function abnormalities (estimated glomerular filtration rate [eGFR] < 60), (4) abdominal aortic aneurysms, and (5) prior coronary artery stent placements or bypass surgery. The study received approval from the Research Ethics Committee of Kaohsiung Chang Gung Memorial Hospital, Taiwan. Written informed consent was obtained from all participants. Initially, 80 patients were enrolled; however, two withdrew for personal reasons, one was excluded due to the discovery of an incidental abdominal aortic aneurysm, and nine were excluded due to prior coronary artery stent placement. Consequently, 68 patients were included in the final analysis.

Patient demographics were reviewed, including age, gender, and the presence of hypertension, diabetes mellitus, lipid profiles (total cholesterol, HDL, and LDL levels from the closest pre-CCTA tests), smoking status, and body mass index (BMI). Hypertension was defined as a history of antihypertensive medication use or resting blood pressure readings of ≥ 140 mmHg systolic or ≥ 90 mmHg diastolic. Diabetes mellitus was defined as a fasting plasma glucose level ≥ 126 mg/dL or prior use of oral hypoglycemic agents or insulin. Smoking status was based on any history of smoking at least one cigarette daily before CCTA.

The data collected were used to assess 10-year atherosclerotic cardiovascular disease (ASCVD) risk, categorized into three groups: low to borderline risk (< 7.4%), intermediate risk (7.5% to 19.9%), and high risk (≥ 20%) according to the guidelines of the American College of Cardiology.

Image Acquisition CCTA and Non-Enhanced Abdominal CT Scan Protocol CCTA was performed using a 640-slice multislice CT scanner (Canon Aquilion One Genesis, Canon Medical Systems, Japan). All participants received sublingual nitroglycerin (0.3 mg) to promote coronary vasodilation prior to imaging. The first phase involved an unenhanced, prospective electrocardiogram (ECG)-gated volume scan for CAC assessment, configured to 120 kVp and 50 mAs with a field of view (FOV) of 16 cm to ensure comprehensive cardiac coverage. Imaging was performed with a rotation time of 0.275 seconds and a slice thickness of 2 mm. Following this, an abdominal aorta scan was performed using a non-ECG-gated sequential scan mode, maintaining identical settings of 120 kVp and 2 mm slice thickness. The inferior aspect of the L5 vertebral body endplate was used as the caudal extent of the abdominal volume to be imaged, covering the iliac bifurcation of the infrarenal abdominal aorta while minimizing radiation exposure to the pelvic genital organs.

For the enhanced CCTA scans, intravenous contrast medium was delivered using a tailored volume of Omnipaque 350 (Iohexol, GE Healthcare, Chicago, IL, USA), calculated at a 1:1 ratio relative to the patient's body weight, capped at a maximum dose of 65 milliliters (mL). Contrast infusion was performed at a rate of 4-5 mL/s, followed by a saline flush of 50 mL at the same rate. Image acquisition was synchronized with the cardiac cycle using automated peak enhancement detection in the ascending aorta, triggering the scan upon reaching a threshold of 100 Hounsfield units (HU), with imaging beginning after a 5-second delay.

The data acquisition protocol was tailored to each patient's heart rate and rhythm. Specifically, a prospectively ECG-triggered volume scan was used to account for heart rates and rhythms, capturing predefined scanning areas during R-R intervals, especially in instances of frequent ectopic beats or irregular heart rates noted during pre-scan ECG monitoring. Imaging system parameters included a gantry rotation time of 0.275 seconds, collimation of 0.5 mm, tube voltage settings ranging from 100 kV to 120 kV, and a tube current-time product between 200 mAs and 450 mAs, with adjustments based on the patient's BMI.

Image Analysis CAC and AAC were quantitatively assessed using the Vitrea workstation (version 7.4.0.462, Vital Images, Plymouth, MN) following the Agatston method. Calcification was identified as a plaque ≥ 1 mm² with a density exceeding a threshold of 130 HU, which was automatically quantified for both AAC and CAC areas. The AAC and CAC scores were calculated by multiplying the area of each region by a weighted score corresponding to the highest density of calcification: 1 for 130-199 HU, 2 for 200-299 HU, 3 for 300-399 HU, and 4 for densities ≥ 400 HU. Three abdominal aortic coverage areas were analyzed, with the aortoiliac bifurcation serving as the caudal boundary (Figure 1). The first coverage (AAC-all) included the entire abdominal aorta from the superior rim of the celiac trunk origin to the aortoiliac bifurcation. The second coverage (AAC-8cm) extended 8 cm cranially from the aortoiliac bifurcation, comprising 40 slices of 2 mm each, while the third coverage (AAC-5cm) extended 5 cm cranially from the aortoiliac bifurcation, comprising 25 slices of 2 mm each.

The CAD-RADS 2.0 classification system was used to assess the severity of coronary stenosis across five distinct categories: CAD-RADS 0 (no visible stenosis, 0% maximal coronary stenosis), CAD-RADS 1 (minimal stenosis, 1-24%), CAD-RADS 2 (mild stenosis, 25-49%), CAD-RADS 3 (moderate stenosis, 50-69%), CAD-RADS 4 (severe stenosis, subdivided into 4A [70-99%] and 4B [left main >50% or three-vessel obstructive disease]), and CAD-RADS 5 (100% occlusion). The plaque burden classification within CAD-RADS 2.0 includes a "P" designation, ranging from P1 to P4, to quantify overall plaque volume. Two assessment methodologies, CAC scoring and the segment involvement score (SIS), were employed: P1 indicated mild plaque burden (CAC of 1-100 or SIS ≤ 2), P2 indicated moderate plaque burden (CAC of 101-300 or SIS 3-4), P3 indicated severe plaque burden (CAC of 301-999 or SIS 5-7), and P4 indicated extensive plaque burden (CAC ≥1000 or SIS ≥8). The most severe classification from these two assessments determined the P subclassification. The study cohort was categorized into two distinct groups based on AAC-all scores of 300, adapted from the CAC score of 300 to differentiate plaque burden into mild to moderate and severe to extensive categories.

The outcome measures in this study were categorized based on the 2022 Coronary Artery Disease-Reporting and Data System (CAD-RADS), which classifies coronary artery stenosis and plaque burden into distinct categories without the use of specific measurement units. Coronary artery stenosis was graded using a numeric scale from 0 to 5, with higher numbers indicating greater severity of stenosis. Plaque volume was categorized using a classification system ranging from P1 to P4, with P4 representing the highest plaque burden.

Statistical Analysis Statistical analysis was performed using SPSS version 22.0 (IBM SPSS, Chicago, IL, USA). Interobserver agreement for CAD-RADS 2.0 was evaluated using Cohen's kappa coefficient, categorized as poor (< 0.20), fair (0.20-0.39), moderate (0.40-0.59), substantial (0.60-0.79), and excellent (≥ 0.80). Prior to analysis, data distribution normality was assessed using the Kolmogorov-Smirnov test. Quantitative data were summarized as mean ± standard deviation or median (interquartile range, IQR) if not normally distributed. A significance level of p < 0.05 was set. Continuous variables were compared using independent t-tests or Mann-Whitney U tests, while chi-square or Fisher's exact tests were applied to categorical variables as appropriate. One-way ANOVA or Kruskal-Wallis one-way ANOVA was used to assess differences in AAC across CAD-RADS categories and plaque burden subclassifications. Spearman correlation analysis was used to examine the relationship between CAC scores and various AAC score coverage areas, with coefficients ranging from very weak to very strong. The effectiveness of different AAC scores was assessed using receiver operating characteristic (ROC) curves to identify optimal cut-offs for predicting CAD-RADS categories and coronary plaque burden, with CAD-RADS categories stratified into groups 0-2 and 3-5, and coronary plaque burden divided into groups P1-P2 (mild to moderate) and P3-P4 (severe to extensive).

ELIGIBILITY:
Inclusion Criteria:

* patients with chest pain or discomfort who were scheduled to undergo cardiac CT for CAC and CCTA
* determined by the treating physician for the evaluation of CAD

Exclusion Criteria:

* severe allergies to contrast agents
* metallic implants in the lumbar spine
* renal function abnormalities (estimated glomerular filtration rate [eGFR] < 60)
* abdominal aortic aneurysms
* prior coronary artery stent placements or bypass surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Image Analysis | From enrollment to the end of treatment at 1 week
  The CAD-RADS 2.0 classification system was used to assess the severity of coronary stenosis across five distinct categories: CAD-RADS 0 (no visible stenosis, 0% maximal coronary stenosis), CAD-RADS 1 (minimal stenosis, 1-24%), CAD-RADS 2 (mild stenosis, 25-49%), CAD-RADS 3 (moderate stenosis, 50-69%), CAD-RADS 4 (severe stenosis, subdivided into 4A [70-99%] and 4B [left main >50% or three-vessel obstructive disease]), and CAD-RADS 5 (100% occlusion).
  The outcome measures in this study were categorized based on the 2022 Coronary Artery Disease-Reporting and Data System (CAD-RADS), which classifies coronary artery stenosis and plaque burden into distinct categories without the use of specific measurement units. Coronary artery stenosis was graded using a numeric scale from 0 to 5, with higher numbers indicating greater severity of stenosis. Plaque volume was categorized using a classification system ranging from P1 to P4, with P4 representing the highest plaque burden.

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Liao, M.D., Study Director — Kaohsiung Chang Gung Memorial Hospital and Chang Gung University College of Medicine, Kaohsiung, Taiwan
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital and Chang Gung University College of Medicine, Kaohsiung, Taiwan, Kaohsiung City, Niao Sung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
If I want to share, I must get the Kaohsiung Chang Gung Memorial Hospital's consent

REFERENCES:
- [Background] Takayama Y, Yasuda Y, Suzuki S, Shibata Y, Tatami Y, Shibata K, Niwa M, Sawai A, Morimoto R, Kato S, Ishii H, Maruyama S, Murohara T. Relationship between abdominal aortic and coronary artery calcification as detected by computed tomography in chronic kidney disease patients. Heart Vessels. 2016 Jul;31(7):1030-7. doi: 10.1007/s00380-015-0712-y. Epub 2015 Jul 12. PMID 26164596
- [Background] Briet M, Burns KD. Chronic kidney disease and vascular remodelling: molecular mechanisms and clinical implications. Clin Sci (Lond). 2012 Oct;123(7):399-416. doi: 10.1042/CS20120074. PMID 22671427
- [Background] van Rosendael AR, van den Hoogen IJ, Gianni U, Ma X, Tantawy SW, Bax AM, Lu Y, Andreini D, Al-Mallah MH, Budoff MJ, Cademartiri F, Chinnaiyan K, Choi JH, Conte E, Marques H, de Araujo Goncalves P, Gottlieb I, Hadamitzky M, Leipsic JA, Maffei E, Pontone G, Shin S, Kim YJ, Lee BK, Chun EJ, Sung JM, Lee SE, Virmani R, Samady H, Sato Y, Stone PH, Berman DS, Narula J, Blankstein R, Min JK, Lin FY, Shaw LJ, Bax JJ, Chang HJ. Association of Statin Treatment With Progression of Coronary Atherosclerotic Plaque Composition. JAMA Cardiol. 2021 Nov 1;6(11):1257-1266. doi: 10.1001/jamacardio.2021.3055. PMID 34406326
- [Background] Schousboe JT, Claflin D, Barrett-Connor E. Association of coronary aortic calcium with abdominal aortic calcium detected on lateral dual energy x-ray absorptiometry spine images. Am J Cardiol. 2009 Aug 1;104(3):299-304. doi: 10.1016/j.amjcard.2009.03.041. Epub 2009 Jun 6. PMID 19616658
- [Background] Williams MC, Earls JP, Hecht H. Quantitative assessment of atherosclerotic plaque, recent progress and current limitations. J Cardiovasc Comput Tomogr. 2022 Mar-Apr;16(2):124-137. doi: 10.1016/j.jcct.2021.07.001. Epub 2021 Jul 16. PMID 34326003
- [Background] Min JK, Shaw LJ, Devereux RB, Okin PM, Weinsaft JW, Russo DJ, Lippolis NJ, Berman DS, Callister TQ. Prognostic value of multidetector coronary computed tomographic angiography for prediction of all-cause mortality. J Am Coll Cardiol. 2007 Sep 18;50(12):1161-70. doi: 10.1016/j.jacc.2007.03.067. Epub 2007 Sep 4. PMID 17868808
- [Background] Williams MC, Newby DE, Dey D, Dweck MR. Response by Williams et al to Letter Regarding Article, "Low-Attenuation Noncalcified Plaque on Coronary Computed Tomography Angiography Predicts Myocardial Infarction: Results From the Multicenter SCOT-HEART Trial (Scottish Computed Tomography of the HEART)". Circulation. 2020 Oct 20;142(16):e244-e245. doi: 10.1161/CIRCULATIONAHA.120.049840. Epub 2020 Oct 19. No abstract available. PMID 33074760
- [Background] Sama C, Abdelhaleem A, Velu D, Ditah Chobufo M, Fongwen NT, Budoff MJ, Roberts M, Balla S, Mills JD, Njim TN, Greathouse M, Zeb I, Hamirani YS. Non-calcified plaque in asymptomatic patients with zero coronary artery calcium score: A systematic review and meta-analysis. J Cardiovasc Comput Tomogr. 2024 Jan-Feb;18(1):43-49. doi: 10.1016/j.jcct.2023.10.002. Epub 2023 Oct 9. PMID 37821352
- [Background] Devia-Rodriguez R, Derksen M, de Groot K, Vedder IR, Zeebregts CJ, Bokkers RPH, Pol RA, de Vries JPM, Schuurmann RCL. Validation of a Length-Adjusted Abdominal Arterial Calcium Score Method for Contrast-Enhanced CT Scans. Diagnostics (Basel). 2023 Jun 1;13(11):1934. doi: 10.3390/diagnostics13111934. PMID 37296786
- [Background] Mori S, Takaya T, Kinugasa M, Ito T, Takamine S, Fujiwara S, Nishii T, Kono AK, Inoue T, Satomi-Kobayashi S, Rikitake Y, Okita Y, Hirata K. Three-dimensional quantification and visualization of aortic calcification by multidetector-row computed tomography: a simple approach using a volume-rendering method. Atherosclerosis. 2015 Apr;239(2):622-8. doi: 10.1016/j.atherosclerosis.2014.12.041. Epub 2014 Dec 24. PMID 25554696
- [Background] Oishi H, Horibe H, Yamase Y, Ueyama C, Takemoto Y, Shigeta T, Hibino T, Kondo T, Suzuki S, Ishii H, Murohara T. Predictive value of abdominal aortic calcification index for mid-term cardiovascular events in patients with acute coronary syndrome. Heart Vessels. 2020 May;35(5):620-629. doi: 10.1007/s00380-019-01527-6. Epub 2019 Nov 9. PMID 31707516
- [Background] Chuang ML, Leslie RW, Massaro JM, Manders ES, Fox CS, Hoffmann U, O'Donnell CJ. Distribution of abdominal aortic calcium by computed tomography: impact of analysis method on quantitative calcium score. Acad Radiol. 2013 Nov;20(11):1422-8. doi: 10.1016/j.acra.2013.08.008. PMID 24119355
- [Background] Agatston AS, Janowitz WR, Hildner FJ, Zusmer NR, Viamonte M Jr, Detrano R. Quantification of coronary artery calcium using ultrafast computed tomography. J Am Coll Cardiol. 1990 Mar 15;15(4):827-32. doi: 10.1016/0735-1097(90)90282-t. PMID 2407762
- [Background] Grundy SM, Stone NJ, Bailey AL, Beam C, Birtcher KK, Blumenthal RS, Braun LT, de Ferranti S, Faiella-Tommasino J, Forman DE, Goldberg R, Heidenreich PA, Hlatky MA, Jones DW, Lloyd-Jones D, Lopez-Pajares N, Ndumele CE, Orringer CE, Peralta CA, Saseen JJ, Smith SC Jr, Sperling L, Virani SS, Yeboah J. 2018 AHA/ACC/AACVPR/AAPA/ABC/ACPM/ADA/AGS/APhA/ASPC/NLA/PCNA Guideline on the Management of Blood Cholesterol: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines. Circulation. 2019 Jun 18;139(25):e1082-e1143. doi: 10.1161/CIR.0000000000000625. Epub 2018 Nov 10. PMID 30586774
- [Background] Goff DC Jr, Lloyd-Jones DM, Bennett G, Coady S, D'Agostino RB, Gibbons R, Greenland P, Lackland DT, Levy D, O'Donnell CJ, Robinson JG, Schwartz JS, Shero ST, Smith SC Jr, Sorlie P, Stone NJ, Wilson PW, Jordan HS, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the assessment of cardiovascular risk: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S49-73. doi: 10.1161/01.cir.0000437741.48606.98. Epub 2013 Nov 12. No abstract available. PMID 24222018
- [Background] O'Connor SD, Graffy PM, Zea R, Pickhardt PJ. Does Nonenhanced CT-based Quantification of Abdominal Aortic Calcification Outperform the Framingham Risk Score in Predicting Cardiovascular Events in Asymptomatic Adults? Radiology. 2019 Jan;290(1):108-115. doi: 10.1148/radiol.2018180562. Epub 2018 Oct 2. PMID 30277443
- [Background] Bastos Goncalves F, Voute MT, Hoeks SE, Chonchol MB, Boersma EE, Stolker RJ, Verhagen HJ. Calcification of the abdominal aorta as an independent predictor of cardiovascular events: a meta-analysis. Heart. 2012 Jul;98(13):988-94. doi: 10.1136/heartjnl-2011-301464. PMID 22668866
- [Background] Skalsky K, Shiyovich A, Hochwald N, Levi A, Zreik L, Tamir S, Shafir G, Briger A, Rahamimov R, Kornowski R, Hamdan A. Coronary Computed Tomography Angiography and Abdominal Aortic Calcification Screening among High-Risk Living Kidney Donors. J Clin Med. 2023 Jul 7;12(13):4541. doi: 10.3390/jcm12134541. PMID 37445576
- [Background] Cury RC, Leipsic J, Abbara S, Achenbach S, Berman D, Bittencourt M, Budoff M, Chinnaiyan K, Choi AD, Ghoshhajra B, Jacobs J, Koweek L, Lesser J, Maroules C, Rubin GD, Rybicki FJ, Shaw LJ, Williams MC, Williamson E, White CS, Villines TC, Blankstein R. CAD-RADS 2.0 - 2022 Coronary Artery Disease-Reporting and Data System: An Expert Consensus Document of the Society of Cardiovascular Computed Tomography (SCCT), the American College of Cardiology (ACC), the American College of Radiology (ACR), and the North America Society of Cardiovascular Imaging (NASCI). J Cardiovasc Comput Tomogr. 2022 Nov-Dec;16(6):536-557. doi: 10.1016/j.jcct.2022.07.002. Epub 2022 Jul 8. PMID 35864070
- [Background] Cury RC, Abbara S, Achenbach S, Agatston A, Berman DS, Budoff MJ, Dill KE, Jacobs JE, Maroules CD, Rubin GD, Rybicki FJ, Schoepf UJ, Shaw LJ, Stillman AE, White CS, Woodard PK, Leipsic JA. CAD-RADS: Coronary Artery Disease - Reporting and Data System: An Expert Consensus Document of the Society of Cardiovascular Computed Tomography (SCCT), the American College of Radiology (ACR) and the North American Society for Cardiovascular Imaging (NASCI). Endorsed by the American College of Cardiology. J Am Coll Radiol. 2016 Dec;13(12 Pt A):1458-1466.e9. doi: 10.1016/j.jacr.2016.04.024. Epub 2016 Jun 15. PMID 27318576
- [Background] Versteylen MO, Kietselaer BL, Dagnelie PC, Joosen IA, Dedic A, Raaijmakers RH, Wildberger JE, Nieman K, Crijns HJ, Niessen WJ, Daemen MJ, Hofstra L. Additive value of semiautomated quantification of coronary artery disease using cardiac computed tomographic angiography to predict future acute coronary syndrome. J Am Coll Cardiol. 2013 Jun 4;61(22):2296-305. doi: 10.1016/j.jacc.2013.02.065. Epub 2013 Apr 3. PMID 23562925
- [Background] Chang HJ, Lin FY, Gebow D, An HY, Andreini D, Bathina R, Baggiano A, Beltrama V, Cerci R, Choi EY, Choi JH, Choi SY, Chung N, Cole J, Doh JH, Ha SJ, Her AY, Kepka C, Kim JY, Kim JW, Kim SW, Kim W, Pontone G, Valeti U, Villines TC, Lu Y, Kumar A, Cho I, Danad I, Han D, Heo R, Lee SE, Lee JH, Park HB, Sung JM, Leflang D, Zullo J, Shaw LJ, Min JK. Selective Referral Using CCTA Versus Direct Referral for Individuals Referred to Invasive Coronary Angiography for Suspected CAD: A Randomized, Controlled, Open-Label Trial. JACC Cardiovasc Imaging. 2019 Jul;12(7 Pt 2):1303-1312. doi: 10.1016/j.jcmg.2018.09.018. Epub 2018 Dec 12. PMID 30553687
- [Background] Mowatt G, Cummins E, Waugh N, Walker S, Cook J, Jia X, Hillis GS, Fraser C. Systematic review of the clinical effectiveness and cost-effectiveness of 64-slice or higher computed tomography angiography as an alternative to invasive coronary angiography in the investigation of coronary artery disease. Health Technol Assess. 2008 May;12(17):iii-iv, ix-143. doi: 10.3310/hta12170. PMID 18462576
- [Background] Ferencik M, Mayrhofer T, Puchner SB, Lu MT, Maurovich-Horvat P, Liu T, Ghemigian K, Kitslaar P, Broersen A, Bamberg F, Truong QA, Schlett CL, Hoffmann U. Computed tomography-based high-risk coronary plaque score to predict acute coronary syndrome among patients with acute chest pain--Results from the ROMICAT II trial. J Cardiovasc Comput Tomogr. 2015 Nov-Dec;9(6):538-45. doi: 10.1016/j.jcct.2015.07.003. Epub 2015 Jul 10. PMID 26229036
- [Background] Motoyama S, Sarai M, Harigaya H, Anno H, Inoue K, Hara T, Naruse H, Ishii J, Hishida H, Wong ND, Virmani R, Kondo T, Ozaki Y, Narula J. Computed tomographic angiography characteristics of atherosclerotic plaques subsequently resulting in acute coronary syndrome. J Am Coll Cardiol. 2009 Jun 30;54(1):49-57. doi: 10.1016/j.jacc.2009.02.068. PMID 19555840
- [Background] Miller JM, Rochitte CE, Dewey M, Arbab-Zadeh A, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic performance of coronary angiography by 64-row CT. N Engl J Med. 2008 Nov 27;359(22):2324-36. doi: 10.1056/NEJMoa0806576. PMID 19038879
- [Background] An C, Lee HJ, Lee HS, Ahn SS, Choi BW, Kim MJ, Chung YE. CT-based abdominal aortic calcification score as a surrogate marker for predicting the presence of asymptomatic coronary artery disease. Eur Radiol. 2014 Oct;24(10):2491-8. doi: 10.1007/s00330-014-3298-3. Epub 2014 Jul 17. PMID 25030461
- [Background] Zweig BM, Sheth M, Simpson S, Al-Mallah MH. Association of abdominal aortic calcium with coronary artery calcium and obstructive coronary artery disease: a pilot study. Int J Cardiovasc Imaging. 2012 Feb;28(2):399-404. doi: 10.1007/s10554-011-9818-1. Epub 2011 Feb 24. PMID 21347596
- [Background] Jurgens PT, Carr JJ, Terry JG, Rana JS, Jacobs DR Jr, Duprez DA. Association of Abdominal Aorta Calcium and Coronary Artery Calcium with Incident Cardiovascular and Coronary Heart Disease Events in Black and White Middle-Aged People: The Coronary Artery Risk Development in Young Adults Study. J Am Heart Assoc. 2021 Dec 21;10(24):e023037. doi: 10.1161/JAHA.121.023037. Epub 2021 Dec 7. PMID 34873926
- [Background] Janjua SA, Massaro JM, Chuang ML, D'Agostino RB, Hoffmann U, O'Donnell CJ. Thresholds for Abdominal Aortic Calcium That Predict Cardiovascular Disease Events in the Framingham Heart Study. JACC Cardiovasc Imaging. 2021 Mar;14(3):695-697. doi: 10.1016/j.jcmg.2020.09.019. Epub 2020 Nov 18. No abstract available. PMID 33221220
- [Background] Kauppila LI, Polak JF, Cupples LA, Hannan MT, Kiel DP, Wilson PW. New indices to classify location, severity and progression of calcific lesions in the abdominal aorta: a 25-year follow-up study. Atherosclerosis. 1997 Jul 25;132(2):245-50. doi: 10.1016/s0021-9150(97)00106-8. PMID 9242971